CLINICAL TRIAL: NCT07037277
Title: An Evaluation of Bemnifosbuvir-Ruzasvir (BEM/RZR) Versus Sofosbuvir-Velpatasvir (SOF/VEL) for the Treatment of Chronic Hepatitis C Virus (HCV) Infection in a Phase 3 Randomized, Controlled, Open-label Study
Brief Title: C-Forward: Efficacy and Safety of BEM/RZR vs SOF/VEL in Subjects With Chronic HCV
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Atea Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AT-01B-008
Record Dates: First submitted 2025-06-10; First posted 2025-06-25 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-09

CONDITIONS: HEPATITIS C VIRUS CHRONIC INFECTION; Hepatitis C, Chronic; Hepatitis C Virus Infection; Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic; Hepatitis C | interventions — sofosbuvir-velpatasvir drug combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bemnifosbuvir - Ruzasvir (BEM/RZR) (Experimental)
  Interventions: Drug: Bemnifosbuvir-Ruzasvir
- Sofosbuvir-Velpatasvir (SOF/VEL) (Active Comparator)
  Interventions: Drug: Sofosbuvir-Velpatasvir

INTERVENTIONS:
Drug: Bemnifosbuvir-Ruzasvir — BEM/RZR Fixed-dose Combination (FDC) tablets administered orally once daily for a total of 8 weeks (in those without cirrhosis) or 12 weeks (in those with compensated cirrhosis)
  Other Names: (BEM/RZR)
  Arms: Bemnifosbuvir - Ruzasvir (BEM/RZR)
Drug: Sofosbuvir-Velpatasvir — SOF/VEL Fixed-dose Combination (FDC) tablets administered orally once daily for a total of 12 weeks
  Other Names: (SOF/VEL)
  Arms: Sofosbuvir-Velpatasvir (SOF/VEL)

SUMMARY:
The purpose of this study is to compare the efficacy and safety of BEM/RZR to SOF/VEL in adults with chronic HCV.

ELIGIBILITY:
Key Inclusion Criteria:

* Use of adequate contraception for females of childbearing potential
* Must be direct-acting antiviral (DAA)-treatment-naïve (never exposed to an approved or experimental DAA for HCV)
* Documented medical history compatible with chronic HCV
* Either no liver cirrhosis or with compensated liver cirrhosis
* If HIV-1-positive, must meet the following 2 criteria:

  1. Antiretroviral (ARV) regimen for >8 weeks prior to screening visit, with CD4 T-cell count >200 cells/mm3 and plasma HIV-1 RNA <LLOQ
  2. Suitable ARV treatment and not taking any contraindicated medications

Key Exclusion Criteria:

* Pregnant or breastfeeding
* Co-infected with hepatitis B virus
* Abuse of alcohol and/or illicit drug use that could interfere with adherence to study requirements as judged by the investigator
* Prior exposure to any HCV DAA
* Requirement of any prohibited medications
* Use of other investigational drugs within 30 days of dosing
* History or signs of decompensated liver disease (decompensated cirrhosis)
* History of hepatocellular carcinoma (HCC)
* Any other clinically significant medical condition that, in the opinion of the investigator, would jeopardize the safety of the subject or impact the validity of the study results

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 880 (Estimated)
Dates: Start 2025-06-02 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Portion of subjects achieving HCV RNA less than the lower limit of quantitation (LLOQ) at week 24 | Day 1 through Week 24

SECONDARY OUTCOMES:
Proportion of subjects achieving HCV RNA < LLOQ 12 weeks after the last dose of study drugs | Day 1 through 12 weeks after the end of treatment
Proportion of subjects experiencing virologic failure as measured by HCV RNA RT-qPCR | Day 1 through Week 24

CONTACTS AND LOCATIONS:
Locations (74):
- France (6):
  - Atea Study Site, Nice, Alpes Maritimes
  - Atea Study Site, Strasbourg, Bas Rhin
  - Atea Study Site, Clichy, Hauts de Seine
  - Atea Study Site, Montpellier, Herault
  - Atea Study Site, Clermont-Ferrand, Puy de Dome
  - Atea Study Site, Créteil, Val de Marne
- Germany (3):
  - Atea Study Site, Hamburg, Hamburg
  - Atea Study Site, Frankfurt am Main, Hesse
  - Atea Study Site, Leipzig, Saxony
- Greece (3):
  - Atea Study Site, Alexandroupoli
  - Atea Study Site, Athens
  - Atea Study Site, Heraklion
- India (16):
  - Atea Study Site, Hyderabad, Andhra Pradesh
  - Atea Study Site, Patna, Bihar
  - Atea Study Site, Rajkot, Gujarat
  - Atea Study Site, Surat, Gujarat
  - Atea Study Site, Shimla, Himachal Pradesh
  - Atea Study Site, Belagavi, Karnataka
  - Atea Study Site, Kochi, Kerala
  - Atea Study Site, Mumbai, Maharashtra
  - Atea Study Site, Nagpur, Maharashtra
  - Atea Study Site, Pune, Maharashtra
  - Atea Study Site, Ludhiana, Punjab
  - Atea Study Site, Agra, Uttar Pradesh
  - Atea Study Site, Kanpur, Uttar Pradesh
  - Atea Study Site, Lucknow, Uttar Pradesh
  - Atea Study Site, Varanasi, Uttar Pradesh
  - Atea Study Site, Kolkata, West Bengal
- Malaysia (5):
  - Atea Study Site, Kota Bharu, Kelantan
  - Atea Study Site, Ampang, Kuala Lumpur
  - Atea Study Site, Kuala Lumpur, Kuala Lumpur
  - Atea Study Site, Kuantan, Pahang
  - Atea Study Site, Kota Kinabalu, Sabah
- Atea Clinical Study Site, Chisinau, Moldova
- Pakistan (5):
  - Atea Study Site, Islamabad
  - Atea Study Site, Karachi
  - Atea Study Site, Lahore
  - Atea Study Site, Peshawar
  - Atea Study Site, Rawalpindi
- Poland (6):
  - Atea Study Site, Krakow
  - Atea Study Site, Kłodzko
  - Atea Study Site, Lublin
  - Atea Study Site, Mysłowice
  - Atea Study Site, Warsaw
  - Atea Study Site, Wroclaw
- Romania (7):
  - Atea Study Site, Bucharest
  - Atea Study Site, Constanța
  - Atea Study Site, Craiova
  - Atea Study Site, Galati
  - Atea Study Site, Iași
  - Atea Study Site, Sibiu
  - Atea Study Site, Suceava
- South Africa (6):
  - Atea Study Site, Port Elizabeth, Eastern Cape
  - Atea Study Site, Bloemfontein, Free State
  - Atea Study Site, Johannesburg, Gauteng
  - Atea Study Site, Pretoria, Gauteng
  - Atea Study Site, Brits, North West
  - Atea Study Site, Somerset West, Western Cape
- South Korea (4):
  - Atea Study Site, Seoul, Gyeonggi-do
  - Atea Study Site, Yangsan, Gyeongsangnam-do
  - Atea Study Site, Busan
  - Atea Study Site, Seoul
- Spain (4):
  - Atea Study Site, Barcelona, Barcelona
  - Atea Study Site, Santander, Cantabria
  - Atea Study Site, Málaga, Malaga
  - Atea Study Site, Vigo, Pontevedra
- Thailand (6):
  - Atea Study Site, Bangkok, Bangkok
  - Atea Study Site, Pathum Wan, Bangkok
  - Atea Study Site, Ratchathewi, Bangkok
  - Atea Study Site, Mueang Nonthaburi, Changwat Khon Kaen
  - Atea Study Site, Hat Yai, Changwat Songkhla
  - Atea Study Site, Mueang Nonthaburi, Chiang Mai
- Turkey (Türkiye) (2):
  - Atea Study Site, Ankara
  - Atea Study Site, Denizli

IPD SHARING:
Plan to Share IPD: Undecided